CLINICAL TRIAL: NCT06112548
Title: The Efficiency of Periarticular Multimodal Drug Injection in Pain Management Following Primary Unilateral Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: The Efficiency of Periarticular Multimodal Drug Injection in Pain Management Following Primary Unilateral TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDMS-Orthopedics-3-2023
Record Dates: First submitted 2023-02-15; First posted 2023-11-01 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Arthritis Knee; Pain; Arthroplasty Complications
Keywords: total knee arthroplasty; arthritis; pain; injection
MeSH Terms: conditions — Pain; Arthritis | interventions — Bupivacaine; Ketorolac; Ketorolac Tromethamine; Epinephrine; Acetaminophen; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TKA with pain management by multimodal periarticular injection. (Experimental): Patients going TKA and getting an injection of a mixture of 20ml of low body weight bupivacaine 5mg/ml plus 1ml of ketorolac 30mg/ml plus 0.5ml adrenaline 1mg/ml injected in medial and lateral retinaculum, medial and lateral collateral ligaments, quadriceps and patellar tendon, joint capsule, subcutaneous fat before closure.
  Interventions: Procedure: primary unilateral TKA; Drug: Bupivacain; Drug: ketorolac; Drug: epinephrine; Drug: Tramadol
- TKA with pain management by IV/oral analgesics. (Experimental): Patients going TKA and getting a standard pain control regime of IV opioids when needed, IV ketorolac, and IV/oral paracetamol.
  Interventions: Procedure: primary unilateral TKA; Drug: Paracetamol; Drug: Ketorolac; Drug: Tramadol

INTERVENTIONS:
Procedure: primary unilateral TKA — Primary unilateral total knee arthroplasty with cruciate scarifying cemented DePuy Synthes PFC Sigma prosthesis.
Drug: Bupivacain — low body weight (0.50%, 20cc) intraoperative periarticular injection
  Arms: TKA with pain management by multimodal periarticular injection.
Drug: ketorolac — 1ml of 30mg/ml ketorolac intraoperative periarticular injection
  Other Names: Toradol
  Arms: TKA with pain management by multimodal periarticular injection.
Drug: epinephrine — 0.5ml Adrenaline 1mg/ml intraoperative periarticular injection
  Other Names: Adrenaline
  Arms: TKA with pain management by multimodal periarticular injection.
Drug: Paracetamol — IV Paracetamol [Ofirmev] introduced every 6 hours after surgery
  Arms: TKA with pain management by IV/oral analgesics.
Drug: Ketorolac — IV Ketorolac {Toradol} introduced every 12 hours after surgery.
  Arms: TKA with pain management by IV/oral analgesics.
Drug: Tramadol — IV Tramadol [Ultram] introduced when needed after surgery

SUMMARY:
This interventional study aims to compare the effectiveness of local multimodal drug periarticular injection in TKA patients with the standard pain control regime that includes opioids, NSAIDs, and other analgesics.

The main questions The investigators strive to answer are:

Is there a significant difference in the severity of pain and functional outcomes when applying periarticular injections? Are there any increased complications when applying the periarticular injections?

DETAILED DESCRIPTION:
The best pain control regime following TKA is controversial. While opioids have an excellent analgesic effect, they also have many side effects. The investigators are conducting a randomized controlled trial to compare the severity of pain following primary unilateral TKA when multimodal drug periarticular injunction is used with the standard pain control regime. The investigators will enroll patients undergoing primary unilateral TKA and randomly allocate them into one treatment group. The first will undergo the procedure with periarticular injection before the closure is composed of a mixture of 20ml of low body weight bupivacaine 5mg/ml plus 1ml of ketorolac 30mg/ml plus 0.5ml adrenaline 1mg/ml injected in medial and lateral retinaculum, medial and lateral collateral ligaments, quadriceps and patellar tendon, joint capsule, subcutaneous fat, and the second will go standard TKA with pain control using opioids, NSAIDS, and paracetamol. The severity of postoperative pain is the primary outcome studied, as well as preoperative complications and any drug side effects, the data will be collected by a fellow researcher who is blinded to the interventions, and the patients will be blinded too. Randomization will be done by a research fellow who is not involved in patient treatment or care.

ELIGIBILITY:
Inclusion Criteria:

* all patients with end-stage arthritis of the knee going primary unilateral total knee arthroplasty.

Exclusion Criteria:

* inflammatory and secondary arthritis of the knee.
* Patients who are allergic to one or more of the drugs used in the injections.
* Patients who are already taking opioids for whatever reason or have a history of addiction.
* BMI less than 20 and more than 35.
* patients with intra-operative complications that would affect the outcomes measurement.
* Patients who are going through complex primary or revision TKA.
* Pregnancy, renal or liver failure.
* Patients who are classified as grade 3 or more according to ASA.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
perception of pain - first assessment | measured 12 hours after surgery.
  The severity of knee pain in the short postoperative period. As stated by the patient, on a scale of 0 to 10, 0 resents no pain at all, and 10 is the worst pain the participant can imagine.
perception of pain - second assessment | measured 24 hours after surgery.
  The severity of knee pain in the short postoperative period. As stated by the patient, on a scale of 0 to 10, 0 resents no pain at all, and 10 is the worst pain the participant can imagine.
perception of pain - third assessment | measured 48 hours after surgery.
  The severity of knee pain in the short postoperative period. As stated by the patient, on a scale of 0 to 10, 0 resents no pain at all, and 10 is the worst pain the participant can imagine.
functional status - first assessment | first measurement four weeks after surgery.
  a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. here, the investigator assesses the function section.
magnitude of disabling pain according to KSS - first assessment | first measurement four weeks after surgery.
  a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100, with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. Here the investigator assesses the pain section.
magnitude of disabling pain according to KSS - second assessment | first measurement six months after surgery.
  a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100, with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. Here the investigator assesses the pain section.
functional status - second assessment | second measurement six months after surgery.
  a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions. here, the investigator assesses the function section.
estimated total blood loss | measured once 48 hours after surgery.
  the total amount of lost blood in the perioperative period and will be calculated using the Gross formula which is estimated by hitting the patients' blood volume by the difference between pre and post-operative hematocrit value divided by the initial hematocrit value

SECONDARY OUTCOMES:
perioperative complications | if happened within 6 months of surgery
  complications such as Venous thromboembolism VTE, infection, drug side effects ETC
opioids consumption - frequency | measured once 48 hours after surgery.
  the amount of consumed opioids measured by times of application in the close postoperative period
opioids consumption - dose | measured once 48 hours after surgery.
  the amount of consumed opioids measured by the dose used in the close postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: jaber ibrahim, MD PHD, Study Chair — Damascus university - faculty of medicine - department of surgery
Locations (1):
- Damascus university, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Mowat F, Ong K, Chan N, Lau E, Halpern M. Prevalence of primary and revision total hip and knee arthroplasty in the United States from 1990 through 2002. J Bone Joint Surg Am. 2005 Jul;87(7):1487-97. doi: 10.2106/JBJS.D.02441. PMID 15995115
- [Background] Hadley S, Day M, Schwarzkopf R, Smith A, Slover J, Zuckerman J. Is Simultaneous Bilateral Total Knee Arthroplasty (BTKA) as Safe as Staged BTKA? Am J Orthop (Belle Mead NJ). 2017 Jul/Aug;46(4):E224-E229. PMID 28856350
- [Background] Lavernia CJ, Alcerro JC, Rossi MD. Fear in arthroplasty surgery: the role of race. Clin Orthop Relat Res. 2010 Feb;468(2):547-54. doi: 10.1007/s11999-009-1101-6. Epub 2009 Sep 18. PMID 19763716
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Shoji H, Solomonow M, Yoshino S, D'Ambrosia R, Dabezies E. Factors affecting postoperative flexion in total knee arthroplasty. Orthopedics. 1990 Jun;13(6):643-9. doi: 10.3928/0147-7447-19900601-08. PMID 2367246
- [Background] Mahoney OM, Noble PC, Davidson J, Tullos HS. The effect of continuous epidural analgesia on postoperative pain, rehabilitation, and duration of hospitalization in total knee arthroplasty. Clin Orthop Relat Res. 1990 Nov;(260):30-7. PMID 1977542
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Sinatra R, Chung KS, Silverman DG, Brull SJ, Chung J, Harrison DM, Donielson D, Weinstock A. An evaluation of morphine and oxymorphone administered via patient-controlled analgesia (PCA) or PCA plus basal infusion in postcesarean-delivery patients. Anesthesiology. 1989 Oct;71(4):502-7. doi: 10.1097/00000542-198910000-00005. PMID 2478049
- [Background] Allen GC, St Amand MA, Lui AC, Johnson DH, Lindsay MP. Postarthroscopy analgesia with intraarticular bupivacaine/morphine. A randomized clinical trial. Anesthesiology. 1993 Sep;79(3):475-80. doi: 10.1097/00000542-199309000-00010. PMID 8363072
- [Background] Smith I, Van Hemelrijck J, White PF, Shively R. Effects of local anesthesia on recovery after outpatient arthroscopy. Anesth Analg. 1991 Nov;73(5):536-9. PMID 1952132
- [Background] Lonner J. Role of liposomal bupivacaine in pain management after total joint arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):37-41. doi: 10.3113/jsoa.2014.0037. PMID 24641895
- [Background] Hendrix JM, Garmon EH. American Society of Anesthesiologists Physical Status Classification System. 2025 Feb 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441940/ PMID 28722969
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034